CLINICAL TRIAL: NCT06547697
Title: EFFECT OF DIFFERENT DIALYSATE SODIUM CONCENTRATIONS ON BLOOD PRESSURE IN CHRONIC HEMODIALYSIS PATIENTS
Brief Title: DIALYSATE SODIUM CONCENTRATION AND BLOOD PRESSURE IN CHRONIC HEMODIALYSIS PATIENTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Principal Investigator, Luka Varda, Assistant, University Medical Centre Maribor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCMaribor
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

ARMS (3):
- Low-to-High (Experimental): In the first period, the participants will be receiving a dialysate sodium concentration of 138 mmol/L, in the second period 140 mmol/L and in the third period 142 mmol/L.
  Interventions: Other: Dialysate sodium concentration
- High-toLow (Experimental): In the first period, the participants will be receiving a dialysate sodium concentration of 142 mmol/L, in the second period 140 mmol/L and in the third period 138 mmol/L.
  Interventions: Other: Dialysate sodium concentration
- No change (Experimental): In all three periods the participants will be recieving the same dialysate sodium concentration of 140 mmol/L.
  Interventions: Other: Dialysate sodium concentration

INTERVENTIONS:
Other: Dialysate sodium concentration

SUMMARY:
While hypertension is one of the most common causes of end-stage renal disease, it is also present in the vast majority of hemodialysis patients. It is associated with higher cardiovascular morbidity and mortality in this group of patients. Altering dialysate sodium concentration presents a possibility of sodium balance control and blood pressure management. However, the ideal dialysate sodium concentration remains a topic for discussion.

Randomised and prospective single dialysis centre study is presented. The participants are randomly divided into 3 groups and will go through 3 periods of 2 months. A "low-to-high" dialysate sodium concentration group will start the study with 138 mmol/L in the first period, continue with 140 mmol/L in the second period and finish with 142 mmol/L. In the "high-to-low" group, the participants will go through the opposite design (reduction from 142 mmol/L to 138 mmol/L over 3 periods). One group will continue with 140 mmol/L throughout the study. Systolic and diastolic BP values before and after dialysis sessions, interdialytic weight gain, ultrafiltration, serum sodium concentration and the presence of hypotension between the groups in each period and within each group over all three periods will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Patients with end-stage renal disease hemodialysis for at least 3 months

Exclusion Criteria:

* Non-cooperation
* Active cancer
* Hospitalization during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2015-03-01 (Actual)

PRIMARY OUTCOMES:
Peridialytic blood pressure | 6 months (3 periods of 2 months)
  Pre- and post dialysis blood pressure values

SECONDARY OUTCOMES:
Interdialytic weight gain | 6 months (3 periods of 2 months)
  Weight gain between dialysis sessions
Ultrafiltration | 6 months (3 periods of 2 months)
  Change of needed ultrafiltration
Serum sodium concentration | 6 months (3 periods of 2 months)
  Change of serum sodium due to the change of dialysate sodium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marshall MR, Wang MY, Vandal AC, Dunlop JL. Low dialysate sodium levels for chronic haemodialysis. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD011204. doi: 10.1002/14651858.CD011204.pub3. PMID 39498822